CLINICAL TRIAL: NCT04988633
Title: "CAP" Fetge Gras. Lifestyle Modification Program of Nurse Management Through a Mobile Application for Patients With MFLD.
Brief Title: "CAP" Fetge Gras. Lifestyle Modification Program in Catalonia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: University of Barcelona (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFG
Record Dates: First submitted 2021-07-22; First posted 2021-08-03 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2021-07

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Liver Diseases; Lifestyle, Healthy
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Phase III, single-centre, randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention CFG App (Experimental): Online healthy lifestyle education through an App. The intervention will consist of viewing educational videos on diet and exercise through an App.
  Interventions: Behavioral: Intervention CFG App
- Control Group (Experimental): Standard tips for healthy lifestyles that are carried out in regular Primary Care practice.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Intervention CFG App — Online healthy lifestyle education through an App. The intervention will consist of viewing educational videos on diet and exercise through an App. Videos will be uploaded to the app on a weekly basis, lasting 2-3.
  Arms: Intervention CFG App
Behavioral: Control Group — Standard tips for healthy lifestyles that are carried out in regular Primary Care practice. After day 1, where standard advice is received, follow-up visits are conducted at week 2, week 4, month 3, and month 6.
  Arms: Control Group

SUMMARY:
The main purpose of this study is to investigate whether an online lifestyle modification program for people with Metabolic Associated Fatty Liver Disease (MAFLD) through a mobile application produces a significant reduction in liver steatosis and is associated with a higher rate of weight loss compared to standard recommendations currently indicated in Primary Care.

DETAILED DESCRIPTION:
Chronic liver disease are very common and potentially severe. For the most part, they are diagnosed in an advanced stage, which prevents the introduction of curative treatments.

MAFLD is currently the most common cause of chronic liver disease affecting approximately 25% of the world's population. MAFLD is characterized by an excessive accumulation of liver fat associated with insulin resistance (IR) which is defined by the presence of steatosis in> 5% of hepatocytes according to histological analysis.

Currently, the only effective strategy for treating MAFLD is weight loss. Several studies show that a 3-5% weight loss manages to reduce hepatic steatosis and associated metabolic parameters. Despite this, a reduction of at least 7-10% is required to improve fibrosis. Guidelines from the European Association for the Study of Liver Diseases (EASL) and the American Association for the Study of Liver Diseases (AASLD) recommend following an energy-restricted diet adjusted to the Mediterranean diet, excluding MAFLD-promoting components (processed products and high in added fructose), and perform physical activity in order to achieve this goal. However, it is a difficult goal to achieve and maintain over time. Epidemiological evidence recommends implementing structured lifestyle modification programs with the goal of losing weight.

In people with MFGNA, participation in structured lifestyle programs may be compromised by work and time constraints. An application-based online intervention may be more appropriate for young people, people of working age, and those living far from primary care. EHealth technology is a possible resource for promoting behavior change but is a little-studied field in lifestyles modification of people with MAFLD. Given the lack of information regarding lifestyle modification programs in people with MAFLD as the main therapeutic intervention in Primary Care (PC), we consider to analyze the effectiveness of an online program based on the Mediterranean diet with calorie restriction, associated with specific goals of weight loss and physical activity, which allows to reduce hepatic steatosis of individuals with MAFLD.

This study, along with studies of early detection of chronic liver disease through liver elastography "LiverScreen", aims to be the beginning of the approach to chronic liver disease in Primary Care. The aim of this study is to evaluate a strategy for treating MAFLD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Fibroscan® with a CAP ≥ 300 dB/m and liver stiffness <8 Kpa.

Exclusion Criteria:

* Serious chronic disease (heart, respiratory, cancer, etc.).
* Chronic liver disease.
* Chronic kidney disease (FGR <60ml/min).
* Weight loss> 5% during the last three months.
* AUDIT- C> 8
* Impossibility to follow the recommended diet (for religious reasons, swallowing problems, etc.) or inability to perform physical activity.
* Inability to follow the scheduled visits to the intervention (institutionalized individuals, lack of autonomy, inability to walk, lack of a stable home, travel plans, etc.).
* Have been included in another weight loss advice program (>5 kg) during the 6 months prior to the selection visit (basal visit).
* History of having followed a low calorie diet (<900Kcal/day) for the last 6 months.
* History of surgical procedures to lose weight or intend to undergo bariatric surgery in the next 12 months.
* Hemoglobin A1c ≥ 9%.
* History of resection of the small or large intestine.
* History of inflammatory bowel disease.
* BMI> 40 or obesity of known endocrine origin (with the exception of treated hypothyroidism).
* Current treatment with systemic corticosteroids.
* Current use of medication for weight loss.
* Current treatment with steatogenic drugs.
* People participating in a clinical trial with drugs.
* Patients with mental incapacity, language barrier, bad social support or any other reason considered by the investigator precluding adequate understanding, cooperation or compliance in the study.
* Refusal to give informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Rate of reduction in hepatic steatosis in people with MAFLD. | Month 12

SECONDARY OUTCOMES:
Liver steatosis improvement rate according to CAP value (dB/m) | Month 6 and 12
Changes from baseline in weight (kg) at month 6 and month 12. | Month 6 and 12
Changes from baseline in abdominal circumference (cm) and anthropometric variables at month 6 and 12. | Month 6 and 12
Adherence to healthy lifestyle with | Month 6 and 12
Changes from baseline in cardiovascular risk through REGICOR at month 6 and 12. | Month 6 and 12
Changes from baseline in lipid profile (TG, total COL, HDL, LDL), glycemia and HbA1c at month 6 and month 12. | Month 6 and 12
Changes from baseline in liver stiffness values for Fibroscan®, FIB-4 and NAFLD-score and on steatosis scores FLI, HSI, ION at month 6 and 12. | Month 6 and 12
Changes from baseline in steatosis scores FLI, HSI, ION at month 6 and 12. | Month 6 and 12
Changes from baseline in quality of life of individuals at month 6 and 12 and throughout the study throught EuroqoL questionnarie. | Month 6 and 12
Satisfaction of individuals in the participation of the study throught adHoc questionnaire | D0, month 6, month 12

CONTACTS AND LOCATIONS:
Locations (1):
- Núria Fabrellas, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No